CLINICAL TRIAL: NCT01150578
Title: Lexi-Echo - a Rapid, Portable, Non-radiating Diagnostic Test for Myocardial Ischemia That is Accurate Relative to Simultaneously Obtained Nuclear SPECT MPI
Brief Title: Evaluation of Myocardial Ischemia Using Standard Single Photon Emission Computed Tomography (SPECT) With Regadenoson and Simultaneous Cardiac Echocardiography
Acronym: Lexi-Echo
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aiden Abidov (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Aiden Abidov, Associate Professor of Medicine and Radiology, University of Arizona
Organization: University of Arizona (Other)
Other Study IDs: Lexi-Echo2010
Record Dates: First submitted 2010-03-09; First posted 2010-06-25 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Myocardial Ischemia
Keywords: Echocardiography, 2D; speckle tracking; Lexiscan; regadenoson; Myocardial ischemia; Myocardial perfusion imaging; cost and cost analysis; Cardiac-Gated SPECT Imaging; Echocardiography
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lexi-Echo pilot: Appropriate patients at University of Arizona Medical Center stress imaging laboratory who have a routine regadenoson SPECT nuclear scan will have simultaneous cardiac echo images obtained.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — No intervention

SUMMARY:
This study is for people who have a SPECT scan (nuclear imaging of the blood flow to the heart muscle) ordered by their medical doctors. As part of the SPECT scan, they will have been given a drug called regadenoson to widen and expand the blood vessels bringing blood to the heart muscle. The SPECT pictures of the heart are taken about an hour after the regadenoson is put into an arm vein through an IV. In this study, additional echo pictures will be taken and compared to the SPECT pictures.

The aim of the study is to see if the echo pictures work as well as SPECT to measure the blood flow to the heart muscle.

DETAILED DESCRIPTION:
This is a single center, prospective, non-randomized, comparative, same-setting study of Lexiscan MPI SPECT versus state-of-the-art echocardiography. Lexiscan SPECT MPI will be performed per routine clinical protocol with Lexiscan administered as per package insert (0.4 mg in 5 ml IV push over 10 seconds followed by a 5 ml saline flush). Simultaneous echo/Doppler will be obtained immediately before (baseline), during and immediately post (peak vasodilation) using conventional techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to a University of Arizona/Sarver Heart Center/University Medical Center stress imaging laboratory and scheduled to receive a regadenoson SPECT nuclear scan.

Exclusion Criteria:

* Patients unable or unwilling to undergo the clinically necessary stress test or to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a University of Arizona / Sarver Heart Center / University Medical Center stress imaging laboratory and scheduled to receive a regadenoson SPECT nuclear scan.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Determine the diagnostic accuracy of state-of-the-art echocardiography after regadenoson administration (Lexi-Echo) in the evaluation of myocardial ischemia (determined by the reference standard myocardial perfusion imaging SPECT). | 10 minutes

SECONDARY OUTCOMES:
Obtain short term (6 month) outcomes: hospitalization for ischemia or infarction, coronary angiographic (invasive or noninvasive) correlation when available for clinical indications, and mortality. | 6 months
Perform a limited cost-analysis of the two diagnostic testing options | 6 months
Obtain hemodynamic Doppler Echo variables to investigate the acute hemodynamic alterations during Lexiscan infusion. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Aiden Abidov, MD, PhD, Principal Investigator — Associate Professor of Medicine and Radiology
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States